CLINICAL TRIAL: NCT03079245
Title: Improving Antimicrobial Prescribing Practices in the Neonatal Intensive Care Unit
Brief Title: Improving Antimicrobial Prescribing Practices in the Neonatal ICU
Acronym: iNAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Weill Medical College of Cornell University (Other); Children's Hospital of Philadelphia (Other); Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Lisa Saiman, Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAC6366; 1R01NR010821-01 (NIH); 1R21NR010823-01 (NIH)
Record Dates: First submitted 2017-03-02; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Infants in Neonatal Intensive Care Units
Keywords: Neonatal ICU; antimicrobial stewardship
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: A pre-post intervention study followed by two years of use of randomly assigned interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NICU A - E+, CDS, and PAF (Other): This site was assigned to three interventions, Education Plus (E+), Clinical Decision Support (CDS), and Prescriber Audit and Feedback (PAB).
  Interventions: Other: Education Plus (E+); Other: Clinical Decision Support; Other: Prescriber Audit and Feedback
- NICU B - E+ and CDS (Other): This site was assigned to two interventions, Education Plus (E+) and Clinical Decision Support (CDS).
  Interventions: Other: Education Plus (E+); Other: Clinical Decision Support
- NICU C - E+ (Other): This site was assigned to one intervention, Education Plus (E+).
  Interventions: Other: Education Plus (E+)
- NICU D - Usual Care (No Intervention): This site was not introduced to an interdisciplinary intervention.

INTERVENTIONS:
Other: Education Plus (E+) — Education Plus was an intervention developed by the study team based on the Center for Disease Control (CDC) 12 Step Campaign to Prevent Antimicrobial Resistance in Healthcare Settings. The study team provided Education Plus quarterly to prescribers at the three sites (NICU A, B, C) randomized to this intervention. Examples of topics presented were an overview of antimicrobial stewardship principles, epidemiology of healthcare-associated infections (HAIs), prevention of surgical site infections, antimicrobial susceptibility testing, and pharmacokinetic principles. Educational formats included didactic lectures, participation via the audience response system, case vignettes, and panel discussions.
  Arms: NICU A - E+, CDS, and PAF; NICU B - E+ and CDS; NICU C - E+
Other: Clinical Decision Support — The CDS tool was an intervention developed in consultation with neonatologists and pediatric infectious disease physicians from NICU A and B. Algorithms for empiric and targeted antimicrobial therapy for common pathogens and common clinical scenarios using local antimicrobial susceptibility patterns were developed. The CDS tool also provided additional components to facilitate antimicrobial prescribing, e.g., patient weight, day of life, previous culture results, antimicrobial orders, and selected laboratory results including white blood cell and platelet count, C-reactive protein, creatinine, and therapeutic drug levels. NICUs A and B also received E+
  Arms: NICU A - E+, CDS, and PAF; NICU B - E+ and CDS
Other: Prescriber Audit and Feedback — The prescriber audit and feedback (PAF) intervention was developed by the study team which held focus groups with neonatologists at NICU A (the site randomized to this intervention) to determine the feedback parameters and feedback format as previously described. Neonatologists at NICU A were provided aggregated prescribing data bimonthly that described inappropriate use as described below and prolonged therapy (>7 days) for culture-negative late onset sepsis. NICU A also received CDS and E+.
  Arms: NICU A - E+, CDS, and PAF

SUMMARY:
To determine if 3 randomly assigned bundles of stewardship interventions would reduce overall and inappropriate antimicrobial use in the neonatal intensive care unit (NICU), a pre-post study was performed in 4 NICUs.

DETAILED DESCRIPTION:
Antimicrobial stewardship can improve the safety and quality of healthcare, reduce antimicrobial resistance, and reduce healthcare costs. However, the optimal strategies for the NICU population are unknown and few studies have evaluated the impact of stewardship in this population. To determine if 3 randomly assigned bundles of stewardship interventions would reduce overall and inappropriate antimicrobial use in the NICU. The investigators hypothesized that the bundle using all three interdisciplinary antimicrobial stewardship strategies (education, computer decision support and prescriber audit and feedback) would more effectively reduce overall and inappropriate antimicrobial use compared to usual care. A pre-post intervention study (one baseline year without interventions - May 1, 2009 - April 30, 2010, followed by two years of interventions - May 1, 2010 - April 30, 2012) was performed in 4 academically affiliated, level III NICUs. The sites were randomly assigned to usual care, one intervention, two interventions, or three interventions.

ELIGIBILITY:
Inclusion Criteria:

* infants admitted to study NICUs <7 days of age who remained hospitalized 4 days or more days

Exclusion Criteria:

* Infants admitted to study NICUs 7 days of age and older who were hospitalized less than 4 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6184 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2012-04-30 (Actual); Study Completion 2012-04-30 (Actual)

PRIMARY OUTCOMES:
Overall Antimicrobial Use measured as days of therapy per 100 patient-days | Through study completion for 2 years
  The indications for initiation of intravenous antimicrobials were categorized as initiation of empiric therapy (antibiotics started prior to culture results), definitive therapy (culture results available prior to initiation of antibiotics), or prophylaxis (e.g., antibiotics for postoperative prophylaxis).

SECONDARY OUTCOMES:
Length of therapy per 100 patient-days | Through study completion for 2 years
  2 agents received on same day counted as one day
Inappropriate Antimicrobial Use | Through study completion for 2 years
  Determined on 4th calendar-day of treatment as redundant therapy and failure to target the pathogen
Number of infants initiated on ineffective empiric therapy | Through study completion for 2 years
  Initiation of ineffective empiric therapy for infants thought to be infected
Proportion of infants treated for culture negative late onset sepsis | Through study completion for 2 years
  The proportion of infants treated for culture negative late onset sepsis lasting more than 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Saiman, MD, MPH, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Christiana Care Health Sciences, Wilmington, Delaware
  - Columbia University Medical Center, New York, New York
  - Weill Cornell University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Larson EL, Patel SJ, Evans D, Saiman L. Feedback as a strategy to change behaviour: the devil is in the details. J Eval Clin Pract. 2013 Apr;19(2):230-4. doi: 10.1111/j.1365-2753.2011.01801.x. Epub 2011 Nov 29. PMID 22128773
- [Result] Patel SJ, Saiman L, Duchon JM, Evans D, Ferng YH, Larson E. Development of an antimicrobial stewardship intervention using a model of actionable feedback. Interdiscip Perspect Infect Dis. 2012;2012:150367. doi: 10.1155/2012/150367. Epub 2012 Feb 21. PMID 22500166
- [Result] Hum RS, Cato K, Sheehan B, Patel S, Duchon J, DeLaMora P, Ferng YH, Graham P, Vawdrey DK, Perlman J, Larson E, Saiman L. Developing clinical decision support within a commercial electronic health record system to improve antimicrobial prescribing in the neonatal ICU. Appl Clin Inform. 2014 Apr 9;5(2):368-87. doi: 10.4338/ACI-2013-09-RA-0069. eCollection 2014. PMID 25024755
- [Result] Prasad PA, Wong-McLoughlin J, Patel S, Coffin SE, Zaoutis TE, Perlman J, DeLaMora P, Alba L, Ferng YH, Saiman L. Surgical site infections in a longitudinal cohort of neonatal intensive care unit patients. J Perinatol. 2016 Apr;36(4):300-5. doi: 10.1038/jp.2015.191. Epub 2015 Dec 10. PMID 26658124
- [Result] Patel SJ, Green N, Clock SA, Paul DA, Perlman JM, Zaoutis T, Ferng YH, Alba L, Jia H, Larson EL, Saiman L. Gram-Negative Bacilli in Infants Hospitalized in The Neonatal Intensive Care Unit. J Pediatric Infect Dis Soc. 2017 Sep 1;6(3):227-230. doi: 10.1093/jpids/piw032. PMID 27302327
- [Result] Clock SA, Ferng YH, Tabibi S, Alba L, Patel SJ, Jia H, DeLaMora P, Perlman JM, Paul DA, Zaoutis T, Larson EL, Saiman L. Colonization With Antimicrobial-Resistant Gram-Negative Bacilli at Neonatal Intensive Care Unit Discharge. J Pediatric Infect Dis Soc. 2017 Sep 1;6(3):219-226. doi: 10.1093/jpids/piw014. PMID 27021036
- [Result] Ferng YH, Clock SA, Wong-Mcloughlin J, DeLaMora PA, Perlman JM, Gray KS, Paul DA, Prasad PA, Zaoutis TE, Alba LR, Whittier S, Larson EL, Saiman L. Multicenter Study of Hand Carriage of Potential Pathogens by Neonatal ICU Healthcare Personnel. J Pediatric Infect Dis Soc. 2015 Sep;4(3):276-9. doi: 10.1093/jpids/piu022. Epub 2014 Mar 30. PMID 26336605